CLINICAL TRIAL: NCT01644318
Title: CXCL9 and CXCL11 Levels in Patients With Autoimmune Thyroiditis and Habitual Abortions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Education and Research Hospital (Other Government)
Other Study IDs: 3848
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Habitual Abortion
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- authoimmıne thyroiditis and habitual abortus
- authoimmune thyroiditis
- healthy controls

SUMMARY:
The purpose of this study is to measure serum CXCL9 and CXCL11 levels in patients with autoimmune thyroiditis and habitual abortions

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women with euthyroid autoimmune thyroiditis and a history of first trimester recurrent spontaneous abortions

Exclusion Criteria:

* 1) presence of acute or chronic systemic diseases; 2) other autoimmune diseases; 3) pregnancy and lactation over the previous 6 months; 4) evidence of infectious diseases in the last 3 months; 5) treatment with drugs known to interfere with cytokine release, such as corticosteroids, immunosuppressors, or nonsteroidal antiinflammatory drugs, amiodarone, and lithium; 6) clinical history of hyperthyroidism and/or the presence of anti-TSH receptor antibodies.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Endocrinology Outpatient Clinic
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Serum CXCL9 and CXCL11 levels in patients with autoimmune thyroiditis and habitual abortions

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Education and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Aktas A, Berberoglu Z, Fidan Y, Yazici AC, Koc G, Aral Y, Ademoglu E, Bekdemir H, Alphan Z. Higher levels of circulating CXCL-9 and CXCL-11 in euthyroid women with autoimmune thyroiditis and recurrent spontaneous abortions. Gynecol Endocrinol. 2014 Feb;30(2):157-60. doi: 10.3109/09513590.2013.871514. Epub 2013 Dec 19. PMID 24351073